CLINICAL TRIAL: NCT00137215
Title: Evaluation of Silverlon Dressing for Autogenous Skin Donor Sites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Institute of Surgical Research (U.S. Federal Agency)
Responsible Party: Leopoldo cancio, COL, MC, USAISR
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-04-018
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2008-07-28 (Estimated); Status verified 2008-07

CONDITIONS: Burns
Keywords: burns; donor site care; Silverlon dressing
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Active Comparator)
  Interventions: Device: Silverlon

INTERVENTIONS:
Device: Silverlon — dressing for donor site mamagement

SUMMARY:
The purpose of this study is to compare one type of dressing against the current standard dressing that is used to cover an unburned area of the skin where a piece of skin is removed to cover another part of the body that was burned.

Hypothesis: The mean healing time for wounds treated with the Silverlon Dressing will be less than the mean healing time for wounds treated with Xeroform Dressing.

DETAILED DESCRIPTION:
At the time of the procedure, donor sites that are symmetrical in size and shape will be selected. Once the grafts have been harvested, the wounds will be randomized for treatment using either the Silverlon dressing or Xeroform. The wound dressings will then be observed at least once a day beginning 72 hours after surgery until healed, defined as 90% or more of the wound surface being confluently re-epithelized.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older; male or female.
* Burn wounds of less than 30% total body surface area (TBSA) with no systemic abnormalities
* Burns do not involve the harvesting area
* Burn wounds require excision and grating of sufficient extent to justify two donor sites of equal and symmetrical size on non-dependent body surface areas
* Scheduled excision and grafting procedures is the first such operation for subject during this hospitalization
* Subject agrees to participate in follow-up evaluations

Exclusion Criteria:

* Critical illnesses requiring ventilator support, systemic infection or hemodynamic instability
* Major acute or chronic illnesses affecting wound healing (e.g. peripheral vascular disease, insulin dependent diabetes, blood clotting disorder)
* Subject receiving medications that inhibit/compromise wound healing (e.g. anticoagulants, antiplatelet drugs, oral steroids). The use of anticoagulants does not include deep vein thrombosis (DVT) prophylaxis.
* Cellulitis or other infection of potential donor site
* Previously harvested donor site
* Subject with greater than 30% TBSA burns
* Subjects with sensitivity to silver or nylon
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-01; Primary Completion 2007-08 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Pain will be less than or equal to with the Silverlon Dressing as compared with Xeroform | 14 days
Cosmetic effect of healing at post operative day 30-45 will be equal to or less than with Silverlon as compared with Xeroform | 30-45 days

SECONDARY OUTCOMES:
Infections associated with donor sites will be equal to or less than with Silverlon as compared with Xeroform | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Albrecht, MD, Principal Investigator — US Army Institute of Surgical Research; Steven E Wolf, MD, Study Director — US Army Institute of Surgical Research
Locations (1):
- US Army Institute of Surgical Research, Fort Sam Houston, Texas, United States

REFERENCES:
- [Background] Bowler PG, Jones SA, Walker M, Parsons D. Microbicidal properties of a silver-containing hydrofiber dressing against a variety of burn wound pathogens. J Burn Care Rehabil. 2004 Mar-Apr;25(2):192-6. doi: 10.1097/01.bcr.0000112331.72232.1b. PMID 15091147